CLINICAL TRIAL: NCT02591849
Title: GLP-1 Restores Altered Insulin and Glucagon Secretion in Post-transplantation Diabetes Mellitus
Brief Title: GLP-1 Effects on Insulin and Glucagon in PTDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Jenssen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2014/666
Record Dates: First submitted 2015-08-17; First posted 2015-10-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Post-transplant Diabetes Mellitus
MeSH Terms: interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucagon-like peptide-1 (GLP-1) (Active Comparator): Twelve eligible renal transplant recipients with PTDM and twelve age, gender, BMI and renal function-matched non-diabetic renal transplant recipients will be randomized to continuous unblinded intravenous infusion of GLP-1 with an infusion rate of 0.8 pmol/kg/min or isotonic saline (placebo) on two experimental days performed 2-4 weeks apart. The GLP-1 infusion will consist of 42.5 nmol/mL GLP-1 (7-36) amide, 12.5 mL 5% human albumin and isotonic saline added to a total volume of 50 mL. After 60 min, a 2 hour hyperglycemic clamp will be initiated, where plasma glucose will be elevated by 5 mmol/L from each individual fasting plasma glucose in both groups. This will be done to measure concentrations of glucagon and insulin in hyperglycemic conditions.
  Interventions: Dietary Supplement: Glucagon-like peptide-1 (GLP-1); Other: Hyperglycemic clamp
- Isotonic saline (Placebo Comparator): The included patients will receive concomitant intravenous infusion of isotonic saline on one of the two experimental days
  Interventions: Other: Isotonic saline; Other: Hyperglycemic clamp

INTERVENTIONS:
Dietary Supplement: Glucagon-like peptide-1 (GLP-1)
  Arms: Glucagon-like peptide-1 (GLP-1)
Other: Isotonic saline
  Arms: Isotonic saline
Other: Hyperglycemic clamp

SUMMARY:
Post-transplantation diabetes mellitus (PTDM) develops in 10-15 % of all renal transplant recipients within 10 weeks after transplantation, and has been associated with increased risk of cardiovascular disease and impaired patient survival. PTDM is primarily believed to be a variant of type 2 diabetes mellitus (T2DM), but the pathophysiology underlying the impaired glucose metabolism in renal transplant recipients with PTDM is unclear and some aspects are still poorly investigated. Hyperglycemic clamp investigations with concomitant infusion of glucagon-like peptide-1 (GLP-1) are warranted for a thorough characterization of the α-cell and β-cell function.

The primary objective of the present study is to investigate whether hyperglucagonemia is present in renal transplant recipients with PTDM. Furthermore, the investigators aim to examine the insulinotropic and glucagon suppressive effects of GLP-1 (compared to placebo) in PTDM patients during fasting glycemia and during hyperglycemic conditions (hyperglycemic clamp), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients more than 1 year post transplant with stable renal function (less than 20% deviation in serum creatinine within the last 2 months) and stable prednisolone dose (maximum 5 mg/day) the last three months before inclusion
* Diagnose of PTDM on standard clinical follow-up performed 8 weeks and 1 year post transplant at OUS-Rikshospitalet (fasting plasma glucose ≥ 7.0 mmol/l and/or 2-hour plasma glucose ≥ 11.1 mmol/l following an oral glucose tolerance test) OR
* Non-diabetic renal transplant recipients with a normal glucose tolerance test (control group)
* > 18 years of age
* BMI 18.5-29.9 kg/m2
* Signed informed consent

Exclusion Criteria:

* Severe liver disease
* Pancreatitis (chronic or acute), previous bowel resection, inflammatory bowel disease, malignancy (previous or actual)
* Estimated GFR < 25 ml/min/1.73 m2
* Pregnant or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Concentration of glucagon during fasting glycemia and during hyperglycemic conditions measured in picomoles per liter | 4 weeks
  The primary objective of the present study is to measure fasting plasma glucagon concentration and the suppression of glucagon during hyperglycemia (hyperglycemic clamp) measured in picomoles per liter with and without concomitant iv infusion of glucagon-like peptide-1 (GLP-1) in renal transplant recipients with and without PTDM

SECONDARY OUTCOMES:
Glucose-potentiated arginine test | 4 weeks
  Investigate the functional reserve capacity in glucagon and insulin release (measurement of functional α-cell and β-cell mass) by a glucose-potentiated arginine test; since arginine is a glucose-independent stimulator of the release of both hormones.
Insulin sensitivity index | 4 weeks
  Estimate insulin sensitivity index (ISI) by recording the glucose infusion rate during the hyperglycemic clamp, corrected for the prevailing plasma insulin concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Halden TA, Egeland EJ, Asberg A, Hartmann A, Midtvedt K, Khiabani HZ, Holst JJ, Knop FK, Hornum M, Feldt-Rasmussen B, Jenssen T. GLP-1 Restores Altered Insulin and Glucagon Secretion in Posttransplantation Diabetes. Diabetes Care. 2016 Apr;39(4):617-24. doi: 10.2337/dc15-2383. Epub 2016 Feb 23. PMID 26908914